CLINICAL TRIAL: NCT04856137
Title: A Phase I/II Study of Relapse/Refractory Diffuse Large B-cell Lymphoma
Brief Title: A Phase I/II Study of Diffuse Large B-cell Lymphoma
Acronym: DLBL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); Shin Kong Wu Huo-Shih Memorial Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1420
Record Dates: First submitted 2019-11-26; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Refractory Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: Phase Ib Dose Escalation
  All patients received:
  Rituximab 375mg/m2 on D1 of each cycle, and Paclitaxel 200mg/m2 on D1 of each cycle, plus, G-CSF 1PC sc qd, starting D7 until ANC recovery Ruxolitinib continuously given (D1-21) in the following dose schema
  Phase II Efficacy Study
  All patients received:
  Rituximab 375mg/m2 on D1 of each cycle, and Paclitaxel 200mg/m2 on D1 of each cycle, plus Ruxolitinib using RP2D daily on D1-21 G-CSF 1PC sc qd, starting D7 until ANC recovery
  Repeat every 21 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): ruxolitinib, paclitaxel, and rituximab
  Interventions: Drug: Rituximab Paclitaxel Ruxolitinib

INTERVENTIONS:
Drug: Rituximab Paclitaxel Ruxolitinib — Rituximab 375mg/m2 on D1 of each cycle Paclitaxel 200mg/m2 on D1 of each cycle Ruxolitinib continuously given (D1-21)
  Other Names: G-CSF 1PC sc qd

SUMMARY:
For continuous variables, mean, median, minimum, and maximum will be used for the descriptive purpose. For categorical variables, frequency and percentage will be used for descriptive statistics. The variables of OS will be estimated by the Kaplan-Meier method. Differences between groups will be calculated using the log-rank test for univariate analysis. Cox's proportional hazards model will be employed to test independent prognostic factors. All calculations will be performed using the Statistical Package of Social Sciences software, version 17.0 (SPSS, Inc., Chicago, IL, USA). The level of statistical significance will be set at 0.05 for all tests.

DETAILED DESCRIPTION:
This is an open-label, single arm, prospective, multiple-center phase Ib/II study.

In phase Ib, a maximum of 18 patients will be enrolled in the dose-finding period to determine the RP2D, dependent on the toxicity of the study drugs. The response rates of salvage chemotherapy regimen in R/R DLBCL were reported to be within the range of 35-65%.3 Assuming that the response rate of traditional salvage therapy has an overall response rate of 35% (H0=0.35) and that our experimental regimen would increase it to 50% (H1=0.50), the estimated sample size according to the Simon's two-stage minimal design will be 49 in the second phase.1 Briefly, among the 31 patients recruited during the first stage, the response should be seen in at least 10 of the cases, the lowest threshold for the trial to be moved into the second stage of the phase II part. Furthermore, for the RPR regimen to be deemed effective, a response must be demonstrated in at least 21 of the whole 49 patients enrolled in the phase II period. This would achieve a power of 80%, with a two-sided type I error rate of 10%. An additional 7 patients will be recruited, for an estimated dropout rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed/refractory CD20+ diffuse large B-cell lymphoma.
2. Age greater than 20 years and younger than 75 years old.
3. Measurable disease
4. Patients must have an ECOG performance status of less than or equal to 2.
5. Patients must have recovered from toxic effects of all prior therapy before entering onto study.
6. A treatment of drug-free interval of at least 3 weeks since the last dose of chemotherapy is required.
7. More than 4 weeks since prior radiotherapy is required.
8. Adequate bone marrow function
9. Adequate renal function with calculated glomerular filtration rate > 15 mL/min
10. Patients must have adequate liver function
11. All patients must sign a document of informed consent indicating their awareness of the investigational nature and the risks of the study.

Exclusion Criteria:

1. Patients who have prior treatment with ruxolitinib or taxane for DLBCL.
2. Pregnant or breast-feeding females.
3. Active or uncontrolled infection.
4. Life expectancy < 6 months
5. Patients with brain or leptomeningeal metastases.
6. Known hypersensitivity to ruxolitinib or paclitaxel
7. Grade III peripheral neuropathy secondary to prior to therapy
8. Second malignancy, except indolent cancers not on active anti-cancer therapy.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 1 year
  The tumor response will be assessed according to IWG Response Criteria.

IPD SHARING:
Plan to Share IPD: No